CLINICAL TRIAL: NCT07224919
Title: AutoFocus360 Sound Quality Preference and Claims Study
Acronym: AF360
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Vaisberg (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Vaisberg, Research Scientist, Sonova AG
Organization: Sonova AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-34243
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participant group (Experimental): Participants will listen to scenes of a talker speaking in two types of noise from either the front, left, rear, and right using AutoFocus360 and fixed directional microphones. Condition order is randomized between participants and masked from participants and experimenters.
  Interventions: Device: AutoFocus 360; Device: Fixed directional microphone

INTERVENTIONS:
Device: AutoFocus 360 — AutoFocus 360 is a feature that enhances speech intelligibility by detecting the direction from where speech is coming from relative to the hearing aid wearer and steering the beamforming towards the direction of the speech.
Device: Fixed directional microphone — Fixed directional microphones delivers static beamforming towards the front of the hearing aid wearer.

SUMMARY:
This study aims to generate clinical evidence to substantiate performance claims for the AutoFocus 360 feature in Sonova hearing aid products. AutoFocus 360 is designed to enhance speech intelligibility by detecting the direction of incoming speech and dynamically steering the beamformer toward the talker, regardless of their position relative to the listener. Preliminary internal testing suggested potential benefits in reducing noise disturbance and improving speech clarity compared to traditional directional microphone modes, with outcomes depending on noise type, talker location, and microphone configuration. The present study will systematically evaluate sound quality and listening performance with AutoFocus 360 versus conventional fixed directional settings to support claims of improved speech understanding in noise.

DETAILED DESCRIPTION:
Claims evidence is required for the AutoFocus 360 feature on upcoming product platforms.

AutoFocus 360 is a feature that enhances speech intelligibility by detecting the direction from where speech is coming from relative to the hearing aid wearer and steering the beamforming towards the direction of the speech. Informal exploratory testing by normal hearing Sonova employees have identified that AutoFocus 360 reduces noise disturbance and improves speech clarity, over other microphones modes with some dependencies on (1) noise type, (2) talker location and (3) specific mode comparisons.

AutoFocus 360 is intended to improve listening by directing the hearing aid beamformer towards the speaker wherever they are relative to the listener (i.e. front, side or rear) compared to other in-noise beamforming, mainly fixed wide directional. Sonova currently does not have any data to support this. Therefore, this study will aim to produce sound quality data showing a benefit for Autofocus 360 over traditional beamforming for the purpose of claim substantiation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-99 years)
* Binaural, symmetric, sensorineural N2 (mild) to N5 (moderate-severe) hearing loss
* Fluent in English

Exclusion Criteria:

* Minors (< 18 years
* Normal hearing or hearing loss > N6 (severe)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Noise disturbance sound quality attribute | During a single 2-hour onsite study session
  Participants will complete an A-B paired-comparison listening task to assess subjective preference for noise disturbance between two hearing aid conditions. During testing, participants will listen to short audio recordings that vary in talker location and noise type. For each trial, participants will indicate which of the two recordings (A or B) has less bothersome background noise. The outcome measure will be the proportion of "A preferred" versus "B preferred" responses aggregated across all trials and participants. Binary preference data will be analyzed using inferential statistics.

SECONDARY OUTCOMES:
Speech clarity sound quality attribute | During a single 2-hour onsite study session
  Participants will complete an A-B paired-comparison listening task to assess subjective preference for speech clarity between two hearing aid conditions. During testing, participants will listen to short audio recordings that vary in talker location and noise type. For each trial, participants will indicate which of the two recordings (A or B) has clearer speech. The outcome measure will be the proportion of "A preferred" versus "B preferred" responses aggregated across all trials and participants. Binary preference data will be analyzed using inferential statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG

IPD SHARING:
Plan to Share IPD: No